CLINICAL TRIAL: NCT05090670
Title: The Impact of Germanium-Embedded Knee Brace on Patient Recovery After Knee Arthroscopy: a Blinded and Randomized Controlled Trial
Brief Title: The Impact of Germanium-Embedded Knee Brace on Patient Recovery After Knee Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Total Sports Medicine & Orthopedics (Other)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IW002
Record Dates: First submitted 2021-10-07; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Knee Arthroscopy; Knee Arthropathy Associated With Other Conditions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Germanium-Embedded Knee Brace (Experimental): Following surgery the patients effected limb would be placed in an Germanium-Embedded Knee Brace
  Interventions: Other: Incrediwear Germanium-Embedded Knee Brace following Knee Arthroscopy
- Replica Knee Brace (Active Comparator): Following surgery the patients effected limb would be placed in a replica knee brace
  Interventions: Other: Replica Knee Brace

INTERVENTIONS:
Other: Incrediwear Germanium-Embedded Knee Brace following Knee Arthroscopy — Germanium-Embedded Knee Brace will be applied to the effected limb following Knee Arthroscopy
  Arms: Germanium-Embedded Knee Brace
Other: Replica Knee Brace — Replica Knee brace will be applied to the effected limb following Knee Arthroscopy
  Arms: Replica Knee Brace

SUMMARY:
Anti-inflammatory brace technology has demonstrated superior clinical outcomes in the management of knee osteoarthritis and accelerate recovery time for Major League Soccer players. Authors have postulated that embedding germanium into cotton garments increases circulation and augments the inflammatory process through a transdermal micro-electromagnetic field. In addition to immunomodulatory effects, knee braces immobilize and stabilize the joint through tactile feedback from the skin. Thus, a germanium-embedded knee brace may provide inflammatory control to augment pain and edema while concomitantly enhancing proprioception. Knee Arthroscopy rehabilitation goals during the acute post-operative phase include diminishment of pain and edema as well as restoration of knee range-of-motion. The presented study intends to assess the impact of a germanium-embedded knee brace on patient recovery after Knee Arthroscopy.

Single-center blinded randomized controlled clinical trial to study effectiveness of germanium-infused knee brace on rehabilitation in patient population undergoing Knee Arthroscopy. Patients will be randomized into germanium-infused knee brace group and compared to a replica knee brace group. Inclusion criteria will include skeletally mature individuals undergoing primary Knee Arthroscopy. Exclusion criteria will include autoimmune disorders and history of surgery on ipsilateral joint. The presented protocol intends to assess the impact of a germanium-embedded knee brace on patient recovery after Knee Arthroscopy. The primary outcome measure was chosen for its implications for the design and conduct of the study,1 including well-validated outcome instrument for comparison, facilitation of a priori power analysis, randomization, and blinding. Secondary outcomes were chosen for their pertinence to surgeon decision-making during patient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years old
* Male or female
* Compliant patient
* BMI less than 35
* Undergoing Knee Arthroscopy within 30 days

Exclusion Criteria:

* Rheumatoid Arthritis
* Poorly controlled diabetes (HgA1c > 7.5)
* Previous blood clots
* BMI greater than 35
* Varicosities on operative leg

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Short Form 36 (SF-36) | 4 weeks
  A well-validated patient reported outcome and the most commonly used outcome instrument in orthopaedics.

SECONDARY OUTCOMES:
Pain Estimation | 6 weeks
  Visual Analog Scale, minimum is 0, maximum is 10 and median is 5
Leg Circumference | 6 weeks
  In centimeters, measure by senior surgeon during physical exam using a tape measure at standard post-operative visits
Knee Range of Motion | 6 weeks
  In degrees, measured by a senior surgeon using a Goniometer, at standard post-operative visits

IPD SHARING:
Plan to Share IPD: No